CLINICAL TRIAL: NCT01235052
Title: Prognostic Evaluation of Fluor 18 Labelled FLUROMISONIDAZOLE (18F-FMISO) Positon Emission Tomography-Computed Tomography (PET-CT) in Head and Neck Squamous Cell Carcinomas
Brief Title: Prognostic Evaluation of 18fmiso Pet-ct in Head and Neck Cancer
Acronym: MISORL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2008/20
Record Dates: First submitted 2009-10-28; First posted 2010-11-05 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2014-08

CONDITIONS: Cancer of Head and Neck; Head and Neck Neoplasms
Keywords: Head and neck neoplasms; Positron Emission Tomography; F18 fluoromisonidazole
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TEP with 18F-FMISO (Experimental): TEP with 18F-FMISO
  Interventions: Radiation: Positon Emission Tomography using 18F-FMISO

INTERVENTIONS:
Radiation: Positon Emission Tomography using 18F-FMISO — We will introduce a pretherapy [18F]-FMISO PET-CT in the treatment planning of patients suffering of head and neck cancer and eligible to a radical treatment with curative intent, consisting of conformational radiotherapy with or without chemotherapy or associated targeted therapy. [18F]-FMISO PET-CT results will not be taken into account for the patients' management. We will test different acquisition protocols and use a wild panel of quantification parameters issued from published studies and originals 'one developed by our team enable to describe [18F]-FMISO uptake. Patients will be followed clinically and para-clinically during two years after the end of the treatment according to the edited recommendations of these tumours type and grade to analyze outcome.

SUMMARY:
Head and neck cancer is the sixth most frequent cancer worldwide, excluding lymphomas and skin cancer. If 18FDG PET is considered today as a standard tool in patients with head and neck squamous cell carcinoma (HNSCC) not only for tumoral or nodal staging but also for assessment of distant metastases and synchronous second primary malignancies, hypoxia is one of the most important prognostic factors in radiotherapy of this type of tumors. The only gold standard method for direct determination of oxygen tension is based on using oxygen electrodes showing a good relation with clinical outcome but complex in its realisation. So, PET using 18F-FMISO has been described to be useful for the non invasive assessment of hypoxia in cancer. Especially in France, the use of this radiotracer is very limited and there is no standardised methodology to acquire and quantify 18F-FMISO signal. So there is a need for a rigorous evaluation of this PET tracer. In another way, it could be a very useful tool for evaluation of new therapies and modification of volumes in radiotherapy.

DETAILED DESCRIPTION:
Hypoxia is one of the major worst prognostic factors of clinical outcome in cancer. It is actually admitted that hypoxia is heterogeneous, variable within different tumour types and that it varies spatially and temporally in a tumor. Hypoxia induce proteomic and gene expression changes that lead to increase angiogenesis, invasion and metastases. So, the hypoxic fraction in solid tumours reduces their sensitivity to conventional treatment modalities, modulating therapeutic response to ionizing radiation or certain chemotherapeutic agents. This is particularly important in head and neck cancers (HNC). Hypoxic cells in solid tumours could influence local failure following radiotherapy and has been associated with malignant progression, loco regional spread and distant metastases and represents an increasing probability of recurrence.

Thus, the non-invasive determination and monitoring of the oxygenation status could be of tumours is of importance to predict patient outcome and eventually modify therapeutic strategies in those tumours. Today, the oxygenation status of individual tumours is not assessed routinely. Numerous different approaches have been proposed to identify hypoxia in tumours. Eppendorf oxygen electrode measurements (pO2 histography) may be considered as a 'gold standard' for hypoxia in human malignancies. However, it is an invasive method being confined to superficial, well accessible tumours and requires many measures. PET using [18F]Fluoro-deoxyglucose (18F-FDG), allows non-invasive imaging of glucose metabolism and takes a growing place in cancer staging, But 18F-FDG can't assess correctly the oxygenation status of tumours. PET with appropriate radiotracers enables non-invasive assessment of presence and distribution of hypoxia in tumours. Nitroimidazoles are a class of electron affinic molecules that were shown to accumulate in hypoxic cells in vitro and in vivo. [18F]-FMISO is the most frequently used tracer ; its intracellular retention is dependent on oxygen tension. Consequently, [18F]-FMISO has been used as a non-invasive technique for detection of hypoxia in humans. Different authors have demonstrated that it is suitable to localize and quantify hypoxia. Thus, [18F]-FMISO PET has been studied to evaluate prognosis and predict treatment response. However, some investigators report an unclear correlation between Eppendorf measurements and standardized uptake values (SUV). This observation may be explained by the structural complexity of hypoxic tumour tissues. Nevertheless, there is a need of standardized procedures to acquire and quantify [18F]-FMISO uptake. Today, the use of this tracer is very limited in clinic and the academic studies have included small populations of patients and suffer of the heterogeneity of technical procedures.

The aim of this study is to determine the optimal acquisition protocol and image reconstruction to describe [18F]-FMISO uptake in HNC, then, to validate [18F]-FMISO-PET as a predictive marker of response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Patients presenting a squamous cell head and neck carcinoma proposed for a radical treatment consisting in conformational radiotherapy with or without chemotherapy or associated targeted therapy
* Signed informed consent

Exclusion Criteria:

* Patients with distant metastases known before inclusion
* Patients suffering of a second cancer or treated before by radiotherapy in the tumour site.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Correlation between a hypoxic volume determined by [18F]-FMISO PET-CT and a treatment response two years after radical treatment. | Inclusion (Day 0) and after two years

SECONDARY OUTCOMES:
Evaluate the potential role of a new biological tumour volume (BTV) taking account hypoxia for the delineation of volumes for radiotherapy treatment planning | Inclusion (Day 0)
Study pathological processes contributing to [18F]-FMISO uptake by the correlation with other parameters considered to be representative of hypoxia in tumours | After two years

CONTACTS AND LOCATIONS:
Overall Officials: CLERMONT-GALLERANDE Henri, MCU-PH, Principal Investigator — University Hospital, Bordeaux; PEREZ Paul, PH, Study Chair — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Hôpital Robert Picqué, Villenave-d'Ornon